CLINICAL TRIAL: NCT06127160
Title: Personalized Antibiotic Treatment in the Emergency Department: Panther Trial
Brief Title: Patient-Directed Antimicrobial Duration in Acute Uncomplicated Pyelonephritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brett A Faine (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor-Investigator, Brett A Faine, Clinical Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202303721
Record Dates: First submitted 2023-10-31; First posted 2023-11-13 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Pyelonephritis Acute
Keywords: cephalexin
MeSH Terms: interventions — Cephalexin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Duration Treatment (Active Comparator)
  Interventions: Drug: Cephalexin
- Patient-directed antimicrobial duration (PDAD) (Experimental)
  Interventions: Drug: Cephalexin or placebo

INTERVENTIONS:
Drug: Cephalexin — Cephalexin 1000 mg by mouth 3 times daily for 10 days
  Arms: Standard Duration Treatment
Drug: Cephalexin or placebo — Cephalexin 1000 mg by mouth 3 times daily for a minimum of 3 days, once participant reports symptom resolution for 24 hours they will switch to placebo for remainder of 10 days of treatment.
  Arms: Patient-directed antimicrobial duration (PDAD)

SUMMARY:
This pilot study will randomize 40 female patients with acute uncomplicated pyelonephritis to receive standard duration of therapy versus patient-directed antimicrobial duration (PDAD). The primary objectives of this pilot trial are to determine the feasibility and safety of conducting a full-scale multi-center randomized controlled trial.

DETAILED DESCRIPTION:
Following informed consent, patients will be randomized to receive 10 days of cephalexin or PDAD (minimum of 3 days of cephalexin followed by placebo once patient reports 24 hours of symptom resolution). Patients will be evaluated at day 1 in-person, then daily using a mobile cellphone application to assess acute uncomplicated pyelonephritis (AUP) symptoms and quality of life (QOL). Urine samples will be collected at in-person visits at day 1, 3 weeks, and 4 weeks. Study feasibility will be assessed through day 90.

ELIGIBILITY:
Inclusion:

* Females between 18 and 55 years of age
* Diagnosis of acute uncomplicated pyelonephritis
* Can be discharged home on oral antimicrobial treatment
* Ability to provide written informed consent in English or Spanish

Exclusion:

* Took antibiotics in the prior 48 hours
* Insulin-dependent diabetes
* End-stage liver disease
* If the patient reports a penicillin allergy, and is deemed to be high-risk using the penicillin allergy clinical decision rule (PEN-FAST)
* Serious allergy (e.g., angioedema, anaphylaxis) to the study medication or a similarly reported allergy to a cephalosporin
* Known or identified hydronephrosis, obstruction, or abscess identified by emergency department ultrasound
* Presence of a kidney stone
* Pregnancy or lactation
* Renal dysfunction (defined as creatinine clearance of less than 30 mL/min)
* Renal transplantation
* Complicated pyelonephritis (defined anatomical or functional abnormality of the urinary tract that predisposes to infection)
* Need for additional antimicrobial therapy for a coexisting infection
* Human immunodeficiency virus (HIV) infection, with either a recent (in the past 6 months) acquired immune deficiency syndrome-defining condition or a cluster of differentiation-4 (CD-4+) T lymphocyte count <200/mm^3

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2024-06-04 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Feasibility of completing all clinical trial activities and follow-up | 90 days
  Percentage of participants that complete all study activities and follow-up through 90 days

SECONDARY OUTCOMES:
Sustained clinical cure | 30 days
  Participant does not require any additional antimicrobial treatment and they do not have a recurrence of symptoms after initial clinical improvement.
Sustained microbiological cure | 30 days
  The bacterial pathogen found at trial entry is sustained to fewer than 1000 CFU/mL.
Clinical and microbiological cure rates after the end of treatment | 15-21 days
  Participant does not require any additional antimicrobial treatment and they do not have a recurrence of symptoms after initial clinical improvement AND the bacterial pathogen found at trial entry is reduced to fewer than 1000 CFU/mL.
Adverse event and side effect event rates | 30 days
Additional health care visits with the chief complaint of urinary tract infection | 30 days
Time to return to normal activities | 30 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Olive View - UCLA Medical Center, Sylmar, California
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa

REFERENCES:
- [Background] Foxman B. The epidemiology of urinary tract infection. Nat Rev Urol. 2010 Dec;7(12):653-60. doi: 10.1038/nrurol.2010.190. PMID 21139641
- [Background] Foxman B. Urinary tract infection syndromes: occurrence, recurrence, bacteriology, risk factors, and disease burden. Infect Dis Clin North Am. 2014 Mar;28(1):1-13. doi: 10.1016/j.idc.2013.09.003. Epub 2013 Dec 8. PMID 24484571
- [Background] Taylor RA, Moore CL, Cheung KH, Brandt C. Predicting urinary tract infections in the emergency department with machine learning. PLoS One. 2018 Mar 7;13(3):e0194085. doi: 10.1371/journal.pone.0194085. eCollection 2018. PMID 29513742
- [Background] Hicks LA, Bartoces MG, Roberts RM, Suda KJ, Hunkler RJ, Taylor TH Jr, Schrag SJ. US outpatient antibiotic prescribing variation according to geography, patient population, and provider specialty in 2011. Clin Infect Dis. 2015 May 1;60(9):1308-16. doi: 10.1093/cid/civ076. Epub 2015 Mar 5. PMID 25747410
- [Background] May L, Cosgrove S, L'Archeveque M, Talan DA, Payne P, Jordan J, Rothman RE. A call to action for antimicrobial stewardship in the emergency department: approaches and strategies. Ann Emerg Med. 2013 Jul;62(1):69-77.e2. doi: 10.1016/j.annemergmed.2012.09.002. Epub 2012 Nov 2. PMID 23122955
- [Background] Flores-Mireles AL, Walker JN, Caparon M, Hultgren SJ. Urinary tract infections: epidemiology, mechanisms of infection and treatment options. Nat Rev Microbiol. 2015 May;13(5):269-84. doi: 10.1038/nrmicro3432. Epub 2015 Apr 8. PMID 25853778
- [Background] Gupta K, Hooton TM, Naber KG, Wullt B, Colgan R, Miller LG, Moran GJ, Nicolle LE, Raz R, Schaeffer AJ, Soper DE; Infectious Diseases Society of America; European Society for Microbiology and Infectious Diseases. International clinical practice guidelines for the treatment of acute uncomplicated cystitis and pyelonephritis in women: A 2010 update by the Infectious Diseases Society of America and the European Society for Microbiology and Infectious Diseases. Clin Infect Dis. 2011 Mar 1;52(5):e103-20. doi: 10.1093/cid/ciq257. PMID 21292654
- [Background] Talan DA, Takhar SS, Krishnadasan A, Abrahamian FM, Mower WR, Moran GJ; EMERGEncy ID Net Study Group. Fluoroquinolone-Resistant and Extended-Spectrum beta-Lactamase-Producing Escherichia coli Infections in Patients with Pyelonephritis, United States(1). Emerg Infect Dis. 2016 Sep;22(9):1594-603. doi: 10.3201/eid2209.160148. PMID 27532362
- [Background] Talan DA, Takhar SS, Krishnadasan A, Mower WR, Pallin DJ, Garg M, Femling J, Rothman RE, Moore JC, Jones AE, Lovecchio F, Jui J, Steele MT, Stubbs AM, Chiang WK, Moran GJ. Emergence of Extended-Spectrum beta-Lactamase Urinary Tract Infections Among Hospitalized Emergency Department Patients in the United States. Ann Emerg Med. 2021 Jan;77(1):32-43. doi: 10.1016/j.annemergmed.2020.08.022. Epub 2020 Oct 31. PMID 33131912
- [Background] Low M, Neuberger A, Hooton TM, Green MS, Raz R, Balicer RD, Almog R. Association between urinary community-acquired fluoroquinolone-resistant Escherichia coli and neighbourhood antibiotic consumption: a population-based case-control study. Lancet Infect Dis. 2019 Apr;19(4):419-428. doi: 10.1016/S1473-3099(18)30676-5. Epub 2019 Mar 4. PMID 30846277
- [Background] Brown KA, Khanafer N, Daneman N, Fisman DN. Meta-analysis of antibiotics and the risk of community-associated Clostridium difficile infection. Antimicrob Agents Chemother. 2013 May;57(5):2326-32. doi: 10.1128/AAC.02176-12. Epub 2013 Mar 11. PMID 23478961
- [Background] McCusker ME, Harris AD, Perencevich E, Roghmann MC. Fluoroquinolone use and Clostridium difficile-associated diarrhea. Emerg Infect Dis. 2003 Jun;9(6):730-3. doi: 10.3201/eid0906.020385. PMID 12781017
- [Background] Sader HS, Biedenbach DJ, Streit JM, Jones RN. Cefdinir activity against contemporary North American isolates from community-acquired urinary tract infections. Int J Antimicrob Agents. 2005 Jan;25(1):89-92. doi: 10.1016/j.ijantimicag.2004.07.006. PMID 15620832
- [Background] Mogle BT, Beccari MV, Steele JM, Fazili T, Kufel WD. Clinical considerations for oral beta-lactams as step-down therapy for Enterobacteriaceae bloodstream infections. Expert Opin Pharmacother. 2019 Jun;20(8):903-907. doi: 10.1080/14656566.2019.1594774. Epub 2019 Mar 25. No abstract available. PMID 30908107
- [Background] Fung-Tomc JC, Huczko E, Stickle T, Minassian B, Kolek B, Denbleyker K, Bonner D, Kessler R. Antibacterial activities of cefprozil compared with those of 13 oral cephems and 3 macrolides. Antimicrob Agents Chemother. 1995 Feb;39(2):533-8. doi: 10.1128/AAC.39.2.533. PMID 7726528
- [Background] Bonsu BK, Shuler L, Sawicki L, Dorst P, Cohen DM. Susceptibility of recent bacterial isolates to cefdinir and selected antibiotics among children with urinary tract infections. Acad Emerg Med. 2006 Jan;13(1):76-81. doi: 10.1197/j.aem.2005.07.032. Epub 2005 Dec 19. PMID 16365328
- [Background] MacGregor RR, Graziani AL. Oral administration of antibiotics: a rational alternative to the parenteral route. Clin Infect Dis. 1997 Mar;24(3):457-67. doi: 10.1093/clinids/24.3.457. PMID 9114201
- [Background] Guay DR. Pharmacodynamics and pharmacokinetics of cefdinir, an oral extended spectrum cephalosporin. Pediatr Infect Dis J. 2000 Dec;19(12 Suppl):S141-6. doi: 10.1097/00006454-200012001-00002. PMID 11144395
- [Background] Kanan M, Atif S, Mohammed F, Balahmar Y, Adawi Y, AlSaleem R, Farhan A, Alghoribi M, Mohammed S, Alshanbari R, Fahad M, Kallab R, Mohammed R, Alassaf D, Hazza A. A Systematic Review on the Clinical Pharmacokinetics of Cephalexin in Healthy and Diseased Populations. Antibiotics (Basel). 2023 Sep 3;12(9):1402. doi: 10.3390/antibiotics12091402. PMID 37760698
- [Background] Leigh AP, Nemeth MA, Keyserling CH, Hotary LH, Tack KJ. Cefdinir versus cefaclor in the treatment of uncomplicated urinary tract infection. Clin Ther. 2000 Jul;22(7):818-25. doi: 10.1016/s0149-2918(00)80054-5. PMID 10945508